CLINICAL TRIAL: NCT04428567
Title: A Pilot Dual-Task Treadmill Training to Improve Gait and Balance in Fragile X-Associated Tremor/Ataxia Syndrome
Brief Title: Treadmill Training in Fragile X-associated Tremor/Ataxia Syndrome
Acronym: FXTAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID 19, the recruitment was halted.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18200205
Record Dates: First submitted 2019-10-01; First posted 2020-06-11 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Fragile X Associated Tremor-ataxia Syndrome
Keywords: Dual-task; feasibility; FXTAS; treadmill training
MeSH Terms: conditions — Fragile X Tremor Ataxia Syndrome | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: The subjects will be randomly assigned to 2 groups: 1) treadmill training group with a cognitive task (Intervention group) 2) Control group. The entire intervention period is 6 weeks in both groups, with interventional training occurring 3 days per week for approximately 45 minutes per session. Evaluations will take place at baseline, 3 weeks, at the end of 6 weeks, and 1 month and 6 months after the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill Exercise + Cognitive Training (Dual-Task) (Experimental): The Dual-Task group will be provided with treadmill training with added simultaneous cognitive training during treadmill exercise training.
  Interventions: Behavioral: Dual-Task Treadmill exercise + Cognitive Training
- Control Group (No Intervention): The control group will be assessed as the intervention group at the same time intervals without the intervention.

INTERVENTIONS:
Behavioral: Dual-Task Treadmill exercise + Cognitive Training — The dual-task regimen will include treadmill exercise of 5-10 min warm-up and cool-down, 30 minutes of running towards target heart rate, combined with respond demands with the addition of cognitive tasks. The level of duration and intensity of treadmill exercise will progressively increase over the duration of 6 weeks.
  Arms: Treadmill Exercise + Cognitive Training (Dual-Task)

SUMMARY:
A pilot trial to determine the feasibility of treadmill training with dual training in patients with Fragile X-Associated Tremor/Ataxia Syndrome (FXTAS).

DETAILED DESCRIPTION:
There is substantial evidence that physical exercise can improve motor and cognitive function in individuals with Parkinson's Disease, traumatic brain injury or chronic stroke survivors. However, to the investigator's knowledge, no studies have explored the effect of treadmill training with or without a cognitive dual Task on gait, balance and cognition in Fragile X - Associated Tremor/Ataxia Syndrome (FXTAS), which is characterized by action tremor, cerebellar gait ataxia, parkinsonism, peripheral neuropathy and cognitive deficits, all of which increase the risk for falls and progressive disability. There are presently no medications or treatment interventions that have been shown to effectively manage the symptoms of FXTAS or delay disease progression, and it is currently not clear whether either the ST or Dual-Task treadmill training paradigms would be feasible or effective in FXTAS.

A total of 10 individuals with FXTAS will recruited from the Rush University Movement Disorders Clinic or the FXTAS Clinic Database at Rush University. The subjects will be assigned to either 6 weeks of dual-task treadmill exercise training combined with a cognitive task (intervention group) occurring 3 times weekly, or control group. The primary outcome measures will be feasibility, safety and patient adherence. The assessments will occur at baseline, week 3, week 6, 1 month & 6 month post-training.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of possible, probable or definite FXTAS
* Able to stand and walk without support for 2 minutes

Exclusion Criteria:

* Any neurologic or musculoskeletal problems
* History of traumatic brain injury
* Significant cardiopulmonary or cardiovascular disease
* Dementia or other significant cognitive impairment
* Unstable psychiatric disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
High levels of program attendance, and retention | 6 weeks
  At each study visit the subjects attend and revisit were taken down throughout the entire intervention period in an attendance/retention log book.
High levels of satisfaction | 6 weeks
  At the end of the entire study a client satisfaction questionnaire was administered and interpreted based on a percent of satisfaction, ranging from zero to one hundred percent, on various satisfactory questions. Zero percent meaning highly unsatisfied and one hundred percent meaning highly satisfied.
High levels of recruitment | 6 months
  Research subjects were recruited using a recruitment flyer for the study and tracked by the number of willing participants.

SECONDARY OUTCOMES:
Change in balance and mobility measured by Instrumented-SWAY (i-SWAY) | 6 weeks
  A test (not a scale) to assess balance and postural sway. Subjects will be asked to stand still with their hands across their chests and their feet positioned a set distance apart (scaled to their height) with a wearable sensor that records movements applied to the lumbar trunk. This sensor will record parameters including mean total sway area, path length, jerk, and sway distance in the mediolateral and anteroposterior directions.
Change in functional mobility measured by Instrumented-WALK (i-WALK) | 6 weeks
  A test to examine fatigue over time and that will also allow more accurate calculation of gait variability indices by increasing the number of steps. The subject will walk 25 meters, turn and walk back, and repeat this until 2 minutes has elapsed.
Change in balance and mobility measured by Mini-BEST balance scale | 6 weeks
  This is a shortened version of the Balance Evaluation systems Test (BESTest). It aims to target and identify 6 different balance control systems and has been used as a performance-based balance measure in many interventions and clinical trials. 1) The original BESTest 4 level (0-3) scoring was revised to 3 levels (0-2) due to redundancy. 2) Total Score = 28 points per test directions. 3) Two items have right and left assessment in which the lower score is used within the total score (directions specify which to use). 4) For research, many studies specify use of both left and right data, thus calculating data based on 32 (vs 28 points).
Change in patient reported confidence in balance measured by Activities-Specific Balance Confidence Scale (ABC) | baseline, week 6, post-training month 1 & month 6
  A 16-item self-report questionnaire in which patients rate their balance confidence for performing activities. Items are rated on a rating scale that ranges from 0 - 100. Score of zero represents no confidence, a score of 100 represents complete confidence. Overall score is calculated by adding item scores and then dividing by the total number of items.
Change in cognitive function measured by the Montreal Cognitive ASsessment (MoCa) | 6 months
  A screening instrument designed to help health professionals detect mild cognitive dysfunction. Subjects will answer questions to measure different areas of cognition including attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal.
Change in cognitive function measured by the Symbol Digit Modalities Test (SDMT) | 6 weeks
  A test for evaluating information processing speed, and the subject uses a reference key to pair specific numbers with given abstract geometric figures in 90 seconds. Scores are the correct number of pairs made in 90 seconds, with greater scores indicating greater cognitive abilities.
Change in cognitive function measured by Controlled Oral Word Association Test (COWAT) | 6 weeks
  A phonemic test for verbal fluency and verbal memory. The COWAT uses the three letter set of C, F, and L to assess phonemic fluency. Subjects will be given 1 min to name as many words as possible beginning with one of the letters.
Change in cognitive function measured by (STROOP) | 6 weeks
  A neuro-psychological test for attention and response inhibition the assess the ability to inhibit cognitive interference while processing a specific stimulus.
Change in cognitive function measured by Digit Span forward and backward test | 6 weeks
  One of the oldest and most widely used test of short-term verbal and working memory. On each trial subjects will be presented with a series of digits appearing one at a time on a computer screen. Subjects will be tested in 2 variants; forward-span and backward-span. In the forward-span, the subject will be asked to recall the digits in the order they appeared. In the backward-span, subjects will be asked to recall the digits in the reverse order they appeared.
Change in health related quality of life measured by the Neuro Quality of Life Survey | 6 months
  Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. It is a self-report of health related quality of life in 17 domains and sub-domains for adults and 11 for children with neurological disorders. Raw scores are converted based on consistent metric (T-distribution) with data from the US general population with a t-score mean of 50 and standard deviation of 10. Adult Banks include 19-45 items. Items are scored on a 5-point scale that uses different language depending on assessment. the questions range from least (1) to most (5) based on frequency of behavior, amount of difficulty, or degree of agreement.
Change in depression measured by the Center for Epidemiologic Studies Depression Scale (CES-D) | 6 weeks
  The CES-D is a brief self-report measure that assesses symptoms of depression in the general population. It is a 20-item, self-report measure designed to be used in the general population that assess current symptoms of depression (i.e. this week). The standard cut-off score suggesting depression >16.
Change in quality of sleep measured by the Pittsburgh Sleep Quality Index (PSQI) questionnaire | 6 weeks
  The PSQI is an effective instrument used to measure the quality and patterns of sleep in adults. it differentiates "poor" from "good" sleep quality by measuring seven different areas over the last month; 19 self-reported items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Five additional questions rated by the respondent's roommate or bed partner are included for clinical purposes and are not scored.
Change in perceived exertion on physical activity intensity measured by the Borg Rating Scale (Borg Rating of Perceived Exertion Scale) | 6 weeks
  The Borg Rating of Perceived Exertion Scale measures physical activity intensity felt by the participant based on the physical sensations a participant experiences during physical activity, including increased heart rate, increased respiration or breathing rate, increased sweating, and muscle fatigue.It is a 20-point scale with verbal descriptors to standardize perceived exertion across tasks and individuals. a score of 0 = nothing at all to 10 = very hard.
Change in physical activity level measured step counts monitored by Fitbit wrist watch | 6 weeks
  The daily steps counts monitored by Fitbit wristband will be used as the measure of physical activity
Change in anxiety measured by the Beck Anxiety Inventory (BAI). | 6 weeks
  The BAI is a self-report measure of anxiety that assesses anxiety symptoms and symptom severity. The BAI can discriminate anxiety from depression. 4-point Likert scale response for anxiety symptoms are severity within a week; the total score is calculated by calculating the sum of 21 items. Minimum score of 0 and a maximum score of 63. Score Interpretation: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Joan A O'Keefe, PhD, PT, Principal Investigator — Rush University Medical Center
Locations (1):
- Kellogg Building 1625 W. Harrison St. Room 235, Chicago, Illinois, United States